CLINICAL TRIAL: NCT03728582
Title: Rehabilitating and Decelerating Language Loss in Primary Progressive Aphasia With Transcranial Direct Current Stimulation (tDCS) Plus Language Therapy
Brief Title: Rehabilitating and Decelerating Language Loss in Primary Progressive Aphasia With tDCS Plus Language Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00174879
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Results first posted 2023-04-19 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Primary Progressive Aphasia; PPA
Keywords: Aphasia; Language therapy; Neurocognitive Disorders; Frontotemporal Dementia; Dementia; Anomia
MeSH Terms: conditions — Aphasia, Primary Progressive; Aphasia; Neurocognitive Disorders; Frontotemporal Dementia; Dementia; Anomia | interventions — Speech Therapy

STUDY DESIGN:
Intervention Model Description: Crossover assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active tDCS plus Speech-Language Therapy (Experimental): Active tDCS will be applied at the beginning of 45min speech-language therapy session and will last for 20 min. Language therapy will be verb naming therapy in a sentence context. This will be followed by sham tDCS plus speech-language therapy after a 2 month washout period.
  Interventions: Device: Active tDCS plus Speech-Language Therapy; Device: Sham tDCS plus Speech-Language Therapy
- Sham plus Speech-Language Therapy (Sham Comparator): Sham tDCS will be applied at the beginning of 45min speech-language therapy session. Language therapy will be oral and written naming. Language therapy will be verb naming therapy in a sentence context. This will be followed by active tDCS plus speech-language therapy after a 2 month washout period.
  Interventions: Device: Active tDCS plus Speech-Language Therapy; Device: Sham tDCS plus Speech-Language Therapy

INTERVENTIONS:
Device: Active tDCS plus Speech-Language Therapy — 1-2 milliamps (mA) of Anodal tDCS stimulation is induced between 5cm X5 cm saline soaked sponges where one sponge is placed on the left inferior frontal gyrus (IFG). The stimulation will be delivered at an intensity of 1-2 mA in a ramp-like fashion for a maximum of 20 minutes. Speech-language therapy will be verb naming therapy in a sentence context.
  Other Names: Active tDCS and speech-therapy
Device: Sham tDCS plus Speech-Language Therapy — Sham tDCS stimulation is provided to the left inferior frontal gyrus (IFG) using a tDCS device. Speech-language therapy will be verb naming therapy in a sentence context.

SUMMARY:
People with Primary Progressive Aphasia (PPA) are is a debilitating disorder characterized by the gradual loss of language functioning, even though cognitive functioning is relatively well preserved until the advanced stages of the disease. There are very few evidence-based treatment options available. This study investigates the behavioral and neural effects of multiple consecutive tDCS sessions paired with language therapy targeting verbs in sentences with individuals with PPA.

DETAILED DESCRIPTION:
Primary Progressive Aphasia (PPA) is a debilitating disorder characterized by the gradual loss of language functioning, even though cognitive functioning is relatively well preserved until the advanced stages of the disease. There are three main PPA variants classified based on the pattern of language impairments and areas of atrophy, but anomia is present across all variants in the earliest stages. While there is a significant amount of research investigating multiple treatment approaches for individuals with aphasia resulting from stroke, individuals with PPA have far fewer treatment options to choose from. Recently, a growing body of literature of treatment in stroke-based aphasia have found promising results for pairing traditional language therapy with non-invasive neurostimulation via transcranial direct current stimulation (tDCS). The small amount of studies of the effects of tDCS applied to left inferior frontal gyrus (IFG) in PPA also yield promising results that show tDCS can enhance generalization to untreated structures. Research in stroke-based aphasia has also shown that language outcomes significantly improve when participants are treated with more complex language stimuli, because this treatment approach results in enhanced generalization. For example, therapy that has participants build sentences around verbs has been found to improve word-level verb and noun naming. The current proposal aims to investigate whether combining the benefits of tDCS while providing verb retrieval therapy that uses sentence building to improve word-level retrieval deficits, will enhance word retrieval deficits in PPA and slow the loss of language functioning. It is hypothesized that Furthermore, the proposed study will investigate the atrophy patterns at baseline, to determine which atrophy patterns are predictive of improved word retrieval. Specifically, this proposal aims: 1) to determine whether tDCS to left IFG coupled with therapy promoting verb retrieval within sentences improve noun and verb retrieval in treated and untreated items in individuals with PPA, and 2) To investigate which patterns of atrophy are predictive of maintenance and generalization of word-retrieval in individuals with PPA following tDCS+therapy vs. sham+therapy. This proposed research will allow the investigators to evaluate the potential benefits and sustainability of tDCS in PPA, the generalization of trained items to untrained items, as well as the deceleration of language loss.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PPA, based on the PPA criteria and presence of naming deficits
* Capable of giving informed consent or indicating another to provide informed consent
* 18 years of age to 100 years of age..

Exclusion Criteria:

* Did not speak English before the age of five
* Less than 10 years of education
* Severe naming deficits
* Significant history of drug or alcohol abuse
* History of psychiatric or neurological problems affecting the brain (besides PPA)
* Has experienced seizures during the previous 12 months
* History of brain surgery or any metal in the head
* Uncorrected visual loss or hearing loss by self-report
* Use of medications that lower the seizure threshold (e.g., methylphenidate) or use of N-Methyl-D-aspartate (NMDA) receptor antagonists (e.g., memantine)
* Scalp sensitivity (per participant report)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shannon M Sheppard, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Active tDCS Plus Speech-Language Therapy First Then Sham Plus Speech-Language Therapy: Active transcranial direct current stimulation (tDCS) will be applied at the beginning of one-hour speech-language therapy session and will last for 20 min. Speech-language therapy provided in 15 one-hour sessions, using verb naming therapy in a sentence context. Therapy is provided 3-5 sessions per week until 15 sessions is reached.This will be followed by sham tDCS plus speech-language therapy after a 2 month washout period.
  Active tDCS plus Speech-Language Therapy: 1-2 milliamp (mA) of Anodal tDCS stimulation is induced between 5cm X5 cm saline soaked sponges where one sponge is placed on the left inferior frontal gyrus (IFG). The stimulation will be delivered at an intensity of 1-2 mA in a ramp-like fashion for a maximum of 20 minutes. Speech-language therapy provided in 15 one-hour sessions, using verb naming therapy in a sentence context.
  Sham tDCS plus Speech-Language Therapy: Sham tDCS stimulation is provided to the left inferior frontal gyrus (IFG) using a tDCS device. Speech-language therapy provided in 15 one-hour sessions, using verb naming therapy in a sentence context.
- Sham Plus Speech-Language Therapy Then Active tDCS Plus Speech-language Therapy: Sham tDCS will be applied at the beginning of one-hour speech-language therapy session. Speech-language therapy provided in 15 one-hour sessions, using verb naming therapy in a sentence context. Therapy is provided 3-5 sessions per week until 15 sessions is reached.This will be followed by active tDCS plus speech-language therapy after a 2 month washout period.
  Sham tDCS plus Speech-Language Therapy: Sham tDCS stimulation is provided to the left inferior frontal gyrus (IFG) using a tDCS device. Speech-language therapy provided in 15 one-hour sessions, using verb naming therapy in a sentence context.
  Active tDCS plus Speech-Language Therapy: 1-2 milliamp (mA) of Anodal tDCS stimulation is induced between 5cm X5 cm saline soaked sponges where one sponge is placed on the left inferior frontal gyrus (IFG). The stimulation will be delivered at an intensity of 1-2 mA in a ramp-like fashion for a maximum of 20 minutes. Speech-language therapy provided in 15 one-hour sessions, using verb naming therapy in a sentence context.
Period: Intervention Period 1 (up to 6 Weeks)
Arm/Group | Active tDCS Plus Speech-Language Therapy First Then Sham Plus Speech-Language Therapy | Sham Plus Speech-Language Therapy Then Active tDCS Plus Speech-language Therapy
Started | 3 | 5
Completed | 3 | 4
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout (8 Weeks)
Arm/Group | Active tDCS Plus Speech-Language Therapy First Then Sham Plus Speech-Language Therapy | Sham Plus Speech-Language Therapy Then Active tDCS Plus Speech-language Therapy
Started | 3 | 4
Completed | 2 | 4
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Intervention Period 2 (Up to 6 Weeks)
Arm/Group | Active tDCS Plus Speech-Language Therapy First Then Sham Plus Speech-Language Therapy | Sham Plus Speech-Language Therapy Then Active tDCS Plus Speech-language Therapy
Started | 2 | 4
Completed | 2 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active tDCS Plus Speech-Language Therapy Versus Sham Plus Speech-Language Therapy: Active tDCS will be applied at the beginning of 45min speech-language therapy session and will last for 20 min. Language therapy will be verb naming therapy in a sentence context. This will be followed by sham tDCS plus speech-language therapy after a 2 month washout period.
  Sham tDCS plus Speech-Language Therapy: Sham tDCS stimulation is provided to the left inferior frontal gyrus (IFG) using a tDCS device. Speech-language therapy will be verb naming therapy in a sentence context.
  Active tDCS plus Speech-Language Therapy: 2 milliamp (mA) of Anodal tDCS stimulation is induced between 5cm X5 cm saline soaked sponges where one sponge is placed on the left inferior frontal gyrus (IFG). The stimulation will be delivered at an intensity of 2 mA in a ramp-like fashion for a maximum of 20 minutes. Sham tDCS will be applied at the beginning of 45min speech-language therapy session. Speech-language therapy will be verb naming therapy in a sentence context.
  Language therapy will be oral and written naming. Language therapy will be verb naming therapy in a sentence context. This will be followed by active tDCS plus speech-language therapy after a 2 month washout period.
Arm/Group | Active tDCS Plus Speech-Language Therapy Versus Sham Plus Speech-Language Therapy
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Accuracy of Naming Trained Verbs (0 to 15, Higher Scores Reflect Better Naming Abilities) as Assessed by Object and Action Naming Battery (OANB)
Description: To determine whether tDCS + language therapy will improve naming performance of participants with Primary Progressive Aphasia more effectively than language therapy alone (the sham condition). The primary outcome variable will be trained verbs on the Object and Action Naming battery (OANBtrained). The OANB has 262 items, scored from 0 to 262, with higher scores on the OANB reflecting better naming abilities. The OANB includes 100 verbs (15 trained, 85 untrained) and 162 nouns.
Time Frame: Baseline, and 4-7 weeks after treatment begins
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS Plus Speech-Language Therapy | Sham Plus Speech-Language Therapy
Number analyzed (Participants) | 7 | 7
score on a scale | 2.3 (.285) | 2.05 (0.15)

2. Secondary Outcome: Change in Accuracy of Naming Untrained Verbs (0 to 85, Higher Scores Reflect Better Naming Abilities) and Nouns (0 to 162, Higher Scores Reflect Better Naming Abilities) as Assessed by Object and Action Naming Battery
Description: To determine whether tDCS + language therapy will improve naming performance of participants with Primary Progressive Aphasia more effectively than language therapy alone (the sham condition). The OANB has 262 items, scored from 0 to 262, with higher scores on the OANB reflecting better naming abilities. There are 100 verbs (15 trained, 85 untrained) on the OANB, and 162 nouns.
Time Frame: Baseline, and 4-7 weeks after treatment begins
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS Plus Speech-Language Therapy | Sham Plus Speech-Language Therapy
Number analyzed (Participants) | 7 | 7
score on a scale | 5.27 (0.43) | -0.408 (0.17)

3. Secondary Outcome: Change in Accuracy of Naming Trained Verbs (0 to 15, Higher Scores Reflect Better Naming Abilities) as Assessed by Object and Action Naming Battery
Description: To determine whether tDCS + language therapy will improve naming performance of participants with Primary Progressive Aphasia more effectively than language therapy alone (the sham condition). The OANB has 262 items, scored from 0 to 262, with higher scores on the OANB reflecting better naming abilities. There are 100 verbs (15 trained, 85 untrained) and 162 nouns on the OANB.
Time Frame: Baseline, and 2 months after treatment ends
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS Plus Speech-Language Therapy | Sham Plus Speech-Language Therapy
Number analyzed (Participants) | 7 | 7
score on a scale | 0.48 (0.12) | 1.0 (0.15)

4. Secondary Outcome: Change in Accuracy of Naming Untrained Verbs (0 to 85, Higher Scores Reflect Better Naming Abilities) and Untrained Nouns (0 to 162, Higher Scores Reflect Better Naming Abilities) as Assessed by Object and Action Naming Battery
Description: as for outcome 2
Time Frame: Baseline, and 2 months after treatment ends
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS Plus Speech-Language Therapy | Sham Plus Speech-Language Therapy
Number analyzed (Participants) | 7 | 7
score on a scale | 4.25 (0.43) | -8.84 (0.09)

5. Secondary Outcome: Change in Functional Communication Skills as Assessed by the Functional Assessment of Communication Skills for Adults (ASHA FACS)
Description: The ASHA FACS will be administered pre-treatment and post-treatment to evaluate changes in functional communication skills. The ASHA FACS is used for measuring the functional communication of adults with speech, language, and cognitive communication disorders. The Communicative Independence Scale will be used, which is rated on a 7-point scale ranging from 1 "does not perform the behavior" to 7 "does perform the behavior". The scores on the Communicative Independence Scale range from a low score of 1 to a high score of 7. A higher score on this subscale indicates better ability to communicate independently.
Time Frame: Baseline, and 4-7 weeks after treatment begins
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS Plus Speech-Language Therapy | Sham Plus Speech-Language Therapy
Number analyzed (Participants) | 7 | 7
score on a scale | 0.215 (0.023) | -0.08 (0.07)

6. Secondary Outcome: Change in Functional Communication Skills as Assessed by the Functional Assessment of Communication Skills for Adults (ASHA FACS)
Description: The ASHA FACS will be administered pre- treatment and post treatment to evaluate changes in functional communication skills. The ASHA FACS is used for measuring the functional communication of adults with speech, language, and cognitive communication disorders. The Communicative Independence Scale will be used, which is rated on a 7-point scale ranging from 1 "does not perform the behavior" to 7 "does perform the behavior". The scores on the Communicative Independence Scale range from a low score of 1 to a high score of 7. A higher score on this subscale indicates better ability to communicate independently.
Time Frame: Baseline, and 2 months after treatment ends
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS Plus Speech-Language Therapy | Sham Plus Speech-Language Therapy
Number analyzed (Participants) | 7 | 7
score on a scale | 0.145 (0.02) | -0.59 (0.03)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Active tDCS Plus Speech-Language Therapy: Active tDCS will be applied at the beginning of 45min speech-language therapy session and will last for 20 min. Language therapy will be verb naming therapy in a sentence context. This will be followed by sham tDCS plus speech-language therapy after a 2 month washout period.
  Active tDCS plus Speech-Language Therapy: 2 milliamp (mA) of Anodal tDCS stimulation is induced between 5cm X5 cm saline soaked sponges where one sponge is placed on the left inferior frontal gyrus (IFG). The stimulation will be delivered at an intensity of 2 mA in a ramp-like fashion for a maximum of 20 minutes. Speech-language therapy will be verb naming therapy in a sentence context.
  Sham tDCS plus Speech-Language Therapy: Sham tDCS stimulation is provided to the left inferior frontal gyrus (IFG) using a tDCS device. Speech-language therapy will be verb naming therapy in a sentence context.
- Sham Plus Speech-Language Therapy: Sham tDCS will be applied at the beginning of 45min speech-language therapy session. Language therapy will be oral and written naming. Language therapy will be verb naming therapy in a sentence context. This will be followed by active tDCS plus speech-language therapy after a 2 month washout period.
  Active tDCS plus Speech-Language Therapy: 2 milliamp (mA) of Anodal tDCS stimulation is induced between 5cm X5 cm saline soaked sponges where one sponge is placed on the left inferior frontal gyrus (IFG). The stimulation will be delivered at an intensity of 2 mA in a ramp-like fashion for a maximum of 20 minutes. Speech-language therapy will be verb naming therapy in a sentence context.
  Sham tDCS plus Speech-Language Therapy: Sham tDCS stimulation is provided to the left inferior frontal gyrus (IFG) using a tDCS device. Speech-language therapy will be verb naming therapy in a sentence context.
Arm/Group | Active tDCS Plus Speech-Language Therapy | Sham Plus Speech-Language Therapy
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active tDCS Plus Speech-Language Therapy (N=7) | Sham Plus Speech-Language Therapy (N=7)
Headache (Nervous system disorders) | 0 (0) | 1 (5) — Headache

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT03728582/Prot_SAP_000.pdf